CLINICAL TRIAL: NCT04649437
Title: Pain Sensitization in Patients With Symptomatic Atrial Fibrillation Compared With Asymptomatic Patients
Brief Title: Atrial Fibrillation Symptoms and Pain Sensitization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Anna Björkenheim, Principal investigator, Region Örebro County
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 274094
Record Dates: First submitted 2020-09-24; First posted 2020-12-02 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Symptoms; Quality of Life; Pain; Conditioning pain modulation; Temporal summation
MeSH Terms: conditions — Atrial Fibrillation; Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symptomatic patients (Other): Subjects with symptoms of atrial fibrillation i.e. AF-6 sum score 30 points or more.
  Interventions: Diagnostic Test: Quantitative sensory testing
- Asymptomatic patients (Other): Subjects with no symptoms of atrial fibrillation i.e. AF-6 sum score = 0.
  Interventions: Diagnostic Test: Quantitative sensory testing

INTERVENTIONS:
Diagnostic Test: Quantitative sensory testing — Quantitative sensory testing recordings will be collected by pressure algometry Assessment of temporal summation of pressure pain and conditioning pain modulation will be used to investigate the involvement of pain sensitization.

SUMMARY:
Atrial fibrillation (AF) is the most common sustained arrhythmia and the number of patients with AF is expected to increase substantially in the coming decades. One third of patients with AF report no AF-associated symptoms, but up to one fourth report severe symptoms such as chest pain. It is well recognized, but unclear why patients' experience of AF-related symptoms, including chest pain, varies so much. Patients with chronic pain show a high degree of central sensitization, i.e. facilitated pain responses to repeated painful stimulation and impaired conditioned pain modulation, compared with controls. It is possible that patients with symptomatic AF may have developed pronounced pain sensitization even in the absence of chest pain as a symptom. No previous study has investigated pain sensitization in patients with AF.

The primary objective is to assess differences in pain sensitization in patients with symptomatic AF compared with patients with asymptomatic AF. Secondary objectives are to study the association of age, sex, AF duration, comorbidities and health-related quality of life to pain sensitization. A total of 30 patients with permanent AF (15 symptomatic and 15 asymptomatic) will be recruited. Patients will complete an AF-specific symptom score and a generic health-related quality of life questionnaire, and physicians will assess AF-related symptoms. Quantitative sensory testing recordings will be collected by pressure algometry. Assessment of temporal summation of pressure pain and conditioning pain modulation will be used to investigate the involvement of pain sensitization.

This preliminary pilot study will be used to estimate sample size for a larger study in which both patients and control subjects will be recruited, to further investigate whether patients with symptomatic AF have increased pain sensitization compared with patients with asymptomatic AF and controls. The studies may have an impact on individualized management of patients with AF in the future.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 20 to 75 years old
* Permanent AF
* Previously completed AF-6
* Written informed consent

Exclusion Criteria:

* Paroxysmal or persistent AF
* Previous pulmonary vein isolation
* Psychiatric or cognitive condition
* Pregnancy
* Previous/current drug or alcohol abuse
* Previous neurological or concomitant musculoskeletal condition
* Continuous analgesic medication

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Differences in pain sensitization | Day 1
  A handheld pressure algometer will be used to assess the pressure pain thresholds over the sternum and the tibialis anterior muscle. Low pressure pain thresholds indicate sensitization. A pin prick will be used to induce temporal summation of pressure pain. Ten consecutive stimuli will be applied over the sternum and tibialis anterior muscle and the patient will be asked to rate the pain intensity on the visual analogue scale (minimum 0, maximum 10, higher scores mean worse pain). Temporal summation of pressure pain will be calculated as the difference in the pain intensity between the first and the last stimulation. High temporal summation of pressure pain scores indicate facilitated temporal summation. The conditioning pain modulation index will be assessed as the increase in pain pressure thresholds during cold pressure test. The lower the difference is, the more sensitization.

SECONDARY OUTCOMES:
Correlation of age, sex, AF duration and comorbidities and HRQoL to pain sensitization | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Department of cardiology, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, statistical analysis plan and informed consent form was shared with Dennis Boye Larsen and Lars Arendt Nielsen in Aalborg, Denmark in a meeting in person in September 2020. The clinical study report and encoded data regarding patient characteristics and results from questionnaires, body charts and quantitative sensory testing was shared with Dennis Boye Larsen and Lars Arendt Nielsen in Aalborg, Denmark, for statistical analysis. Data was made available by an encrypted usb flash drive sent by post. There is no other plan to make individual participant data available to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The encoded individual participant data is available for Dennis Boye Larsen and Lars Arendt Nielsen from 14th January 2021 to the end of march 2021.

REFERENCES:
- [Derived] Jackson A, Frobert O, Boye Larsen D, Arendt-Nielsen L, Bjorkenheim A. Patients with symptomatic permanent atrial fibrillation show quantitative signs of pain sensitisation. Open Heart. 2021 Jun;8(1):e001699. doi: 10.1136/openhrt-2021-001699. PMID 34140311

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT04649437/Prot_SAP_000.pdf